CLINICAL TRIAL: NCT03467360
Title: Phase I Trial of CArbonic Anhydrase Inhibition in Combination With Radiochemotherapy or Radioimmunotherapy in Small Cell Lung Carcinoma
Acronym: ICAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/14; 2022-503093-36-00 (EU CTIS Number); 2017-002160-40 (EudraCT Number)
Record Dates: First submitted 2018-01-18; First posted 2018-03-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer
Keywords: acetazolamide
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Acetazolamide; Platinum; Radioimmunotherapy

STUDY DESIGN:
Intervention Model Description: Phase I study with a prospective, multicenter, non randomized, open-label extension cohort, evaluating the safety of acetazolamide in combination with platinum and etoposide-based radiochemotherapy in patients with Localized Small cell lung cancer or in combinaison with radioimmunotherapy in patients with extensive Small cell lung cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Localized SCLC (Experimental): non randomized, open-label extension cohort, evaluating the safety of acetazolamide in combination with platinum and etoposide-based radiochemotherapy in patients with Localized small lung cancer
  Interventions: Drug: acetazolamide in combination with platinum and etoposide-based radiochemotherapy
- Extensive SCLC (Other): non randomized, open-label extension cohort, evaluating the safety of acetazolamide in combination with radioimmunotherapy in patients with extensive small cell lung cancer
  Interventions: Drug: acetazolamide in combination with radioimmunotherapy in patients with extensive SCLC

INTERVENTIONS:
Drug: acetazolamide in combination with platinum and etoposide-based radiochemotherapy — Radiation therapy will be combined with platinum and etoposide-based chemotherapy combined with 3-6 tablets per day of acetazolamide during the entire course of therapy (dosage appropriate to the inclusion phase).
  Arms: Localized SCLC
Drug: acetazolamide in combination with radioimmunotherapy in patients with extensive SCLC — acetazolamide in combination with radioimmunotherapy in patients with extensive SCLC
  Arms: Extensive SCLC

SUMMARY:
The investigators propose to study the carbonic anhydrase inhibition (acetazolamide) associated with concomitant radiochemotherapy or radioimmunotherapy in small cell lung cancer due to:

1. The over-expression of carbonic anhydrases in this type of cancer,
2. The Anti-tumor effect in preclinical acetazolamide in various tumor lines including neuroendocrine tumor lines,
3. The observed synergy between irradiation and inhibition of carbonic anhydrases,
4. Potential anti-tumor immune effect caused by decreased extracellular acidity.

DETAILED DESCRIPTION:
Compared with healthy cells, glucose metabolism is greatly modified in cancer cells because of their highly proliferative character. This differential tumor / healthy tissue property is an opportunity to be able to propose a treatment whose therapeutic gain can be major (targeted treatment). Preclinical studies are multiple and showed that the targeting of overexpressed proteins (carbonic anhydrases) and involved in glycolytic metabolism can lead to a significant anti-tumor effect. This has never been tested in humans.

Acetazolamide is a molecule commonly used for non carcinologic purposes but has demonstrated anti-tumor activity in preclinical studies; there is also synergy radiotherapy / targeting of carbonic anhydrases. Therefore, the investigators propose to study the combination of acetazolamide / radiotherapy / chemotherapy with platinum and etoposide in localized Small Cell Lung cancer, or associated with radioimmunotherapy (extensive SCLC).

This would be the first study:

* targeting glucose metabolism,
* testing the effectiveness of acetazolamide in oncology,
* testing the synergy radiotherapy / targeting glycolytic metabolism,
* trying to manipulate the anti-tumor immune system indirectly, by decreasing extracellular acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years,
* Performance Status 0 to 2,
* Patient with an histologically non-metastatic localized (or extensive SCLC sub-group) Small cell lung cancer,
* Patient who must start radiotherapy treatment combined with chemotherapy with platinum and etoposide (localized SCLC sub-group) or Patient who received 4 cycles of chemoimmunotherapy with platinum salts, etoposide and immunotherapy (atezolizumab or durvalumab) as the first treatment (extensive SCLC sub-group) Note: The decision of the Multidisciplinary Consultation Team must be notified in the patient's medical file,
* Evaluation lesion according to the criteria RECIST 1.1 and / or according to the criteria PERCIST 1.0,
* Women of childbearing potential must have a negative serum pregnancy test within 72 hours of the first administration of the study treatment,
* If the patient is a woman of childbearing potential, she must be surgically sterile or agree to use two adequate methods of contraception throughout the duration of the study until 1 month after the last administration of the study treatment. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year, Note: Abstinence is acceptable if it is the patient's usual and preferred form of contraception,
* If the male patient has one or more female partners of childbearing age, he / she must agree to use an adequate method of contraception, starting at the first administration of the study treatment up to 1 month after the last administration of the treatment. of the study, Note: Abstinence is acceptable if it is the patient's usual and preferred form of contraception,
* Patient willing and able to provide written informed consent/assent for the trial,
* Patient affiliated with a health insurance system.

Exclusion Criteria:

* Patient with metastatic disease,
* History of thoracic irradiation or near / in the thoracic irradiation field,
* Patient who refuses to participate in the study or unable to agree,
* Contraindication to thoracic radiotherapy treatment: congestive heart failure unbalanced (ejection fraction <30%, clinical signs), severe respiratory failure:

  * COPD grade IV according to the GOLD classification,
  * Some GOLD III COPD and any patient with a respiratory defect defined as: oxygen dependence and / or FEV1 <40% normal and / or, DLCO <40% predictive value and / or vital capacity <40% predictive value,
* Contraindication to acetazolamide: hypersensitivity to acetazolamide, severe hepatic, renal or adrenal insufficiency, sulfonamide intolerance, history of renal colic, allergy to wheat other than celiac disease,
* Patient currently receiving one or more treatments described in section 6.9 of the protocol,
* History of cancer, with the exception of cancers in complete remission for more than 5 years, completely resected basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer,
* People particularly vulnerable as defined in Articles L.1121-5 to -8 of the French Healthcare Code, including: person deprived of freedom by an administrative or judicial decision, adult being the object of a legal protection measure or outside a state to express their consent, pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2027-04-27 (Estimated)

PRIMARY OUTCOMES:
To identify the Tolerated Maximum Dose (DMT) and Recommended Dose (DR) of acetazolamide in combination with radiotherapy combined with platinum and etoposide chemotherapy (localized SCLC) or with radioimmunotherapy (extensive SCLC) | 8 months
  The frequency of limiting dose toxicities determined by the number of Adverse Events as Assessed by CTCAE v4.03 :
  * during the 6 weeks of treatment with acetazolamide / chemoradiation based on platinum and etoposide and in the first 6 months of follow-up after the last administration of the treatment
  * during the 10 days of treatment with acetazolamide / radioimmunotherapy and in the first 6 months after the last administration of the treatment with radioimmunotherapy, for the "extensive SCLC" subgroup

SECONDARY OUTCOMES:
To determine the overall tolerance of the association acetazolamide and radiochemotherapy (localized SCLC) or of the association acetazolamide and radioimmunotherapy (extensive)SCLC) | 27 months
  The overall tolerability of the treatments will be measured by clinical (performance status), laboratory (blood sample), and paraclinical evaluations (ETT, EFR) and defined on the NCI CTCAE V4.03 scale
To evaluate the effectiveness of the treatment | 24 months
  The tumor response (complete or partial, stabilization, progression) will be performed by Morphological evaluations using a scanner according to RECIST 1.1 criteria
To evaluate the effectiveness of the treatment | 24 months
  The tumor response (complete or partial, stabilization, progression) will be performed by Metabolic evaluations using a PET-CT scan according to the criteria PERCIST 1.0
To identify predictive factors for response to acetazolamide | 3 months
  The evaluation of predictive factors of acetazolamide response will be determined by serum CAIX and CAXII levels (in the 7 days before the start of acetazolamide and the end-of-treatment visit)
To identify predictive factors for response to acetazolamide | 30 months
  The evaluation of predictive factors of acetazolamide response will be determined by:
  o The initial 18-FDG PET-CT scan (SUVmax, SULpeak) fixation intensity and 3 months after treatment,
To evaluate progression-free survival at 24 months | 24 months
  To determine the delay between the date of inclusion and the date of progression or death
To evaluate overall survival at 24 months | 24 months
  To determine the delay between the date of inclusion and the date of death
To determine the compliance of acetazolamide | 27 months
  Compliance assessment will be done using Girerd's questionnaire
To evaluate the quality of life | 27 months
  Quality of life will be determined using EORTC QLQC30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa VIDAL, Study Director — Centre Antoine Lacassagne
Locations (2):
- Centre Antoine Lacassagne, Nice, France
- Centre Hospitalier Princesse grace, Monte Carlo, Monaco

IPD SHARING:
Plan to Share IPD: No